CLINICAL TRIAL: NCT04627532
Title: A PHASE 1, RANDOMIZED, DOUBLE-BLIND, SPONSOR-OPEN, PLACEBO CONTROLLED, DOSE ESCALATION STUDY TO EVALUATE THE SAFETY, TOLERABILITY, AND PHARMACOKINETICS OF SINGLE ASCENDING DOSES OF PF-07304814 ADMINISTERED AS A 24-H IV INFUSION IN HEALTHY ADULT PARTICIPANTS
Brief Title: Single Ascending Dose Study of Intravenous Infusion of PF 07304814 in Healthy Adult Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: C4611007
Record Dates: First submitted 2020-10-21; First posted 2020-11-13 (Actual); Last update posted 2021-01-06 (Actual); Status verified 2020-12

CONDITIONS: Healthy
Keywords: SAD, Healthy
MeSH Terms: interventions — lufotrelvir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment (Experimental): PF-07304814 assignment
  Interventions: Drug: PF-07304814
- Placebo (Placebo Comparator): Placebo assigned
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PF-07304814 — Participants will receive PF-07304814
  Arms: Treatment
Drug: Placebo — Participants will recieve placebo
  Arms: Placebo

SUMMARY:
The current study is the second clinical administration with PF-07304814, the phosphate prodrug of the active moiety PF-00835231, and the first in healthy adult participants. It is to evaluate safety, tolerability and PK of single escalating doses of PF 07304814 given as a 24-h IV infusion.

DETAILED DESCRIPTION:
The current study is the second clinical administration with PF-07304814, the phosphate prodrug of the active moiety PF-00835231, and the first in healthy adult participants. It is to evaluate safety, tolerability and PK of single escalating doses of PF 07304814 given as a 24-h IV infusion. This is a randomized, double-blind, sponsor-open, placebo-controlled trial. There will be 2 cohorts with a total of approximately 16 participants planned (approximately 8 participants in each cohort).

ELIGIBILITY:
Inclusion Criteria:

* Male and female participants must be 18 to 60 years of age. All fertile participants must agree to use a highly effective method of contraception.
* Male and female participants who are overtly healthy as determined by medical evaluation including medical history, physical examination.
* Participants who are willing and able to comply with all scheduled visits, treatment plan, laboratory tests, lifestyle considerations, and other study procedures.

BMI of 17.5 to 30.5 kg/m2; and a total body weight >50 kg (110 lb).

* Capable of giving signed informed consent.

Exclusion Criteria

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurological, or allergic disease.
* History of HIV infection, hepatitis B, or hepatitis C; positive testing for HIV, HBsAg, or HCVAb. Hepatitis B vaccination is allowed.
* Other medical or psychiatric condition including recent (within the past year) or active suicidal ideation/behavior or laboratory abnormality that may increase the risk of study participation.
* History of venous thromboembolic event, including deep venous thrombosis or pulmonary embolism.
* Use of prescription or nonprescription drugs and dietary and herbal supplements within 7 days or 5 half lives (whichever is longer) prior to the first dose of study intervention
* Previous administration with an investigational drug within 30 days (or as determined by the local requirement) or 5 half-lives preceding the first dose of study intervention used in this study (whichever is longer).
* A positive urine drug test at screening or admission and confirmed by repeat test, if deemed necessary.
* Screening supine BP ≥140 mm Hg (systolic) or ≥90 mm Hg (diastolic), following at least 5 minutes of supine rest.
* Baseline 12 lead ECG that demonstrates clinically relevant abnormalities that may affect participant safety or interpretation of study results
* History of alcohol abuse or binge drinking and/or any other illicit drug use or dependence within 6 months of Screening.
* Blood donation (excluding plasma donations) of approximately 1 pint (500 mL) or more within 60 days prior to dosing.
* Investigator site staff or Pfizer employees directly involved in the conduct of the study, site staff otherwise supervised by the investigator, and their respective family members

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2020-10-23 (Actual); Primary Completion 2020-12-17 (Actual); Study Completion 2020-12-17 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment emergent treatment-related adverse event(s) | Dosing through follow-up call (28-32 days after last dose of investigational product)
  Frequency, severity and causal relationship of treatment emergent adverse events (TEAEs) and withdrawals due to TEAEs
Number of participants with laboratory test findings of potential clinical importance | Dosing through Day 5 of last period
  Percentage of subjects with laboratory abnormalities
Number of participants with vital signs findings of potential clinical importance | Dosing through Day 5 of last period
  blood pressure, pulse rate, temperature, respiration rate
Number of participants with ECG findings of potential clinical importance | Dosing through Day 5 of last period
  Number of subjects with change from baseline in electrocardiogram (ECG) parameters

SECONDARY OUTCOMES:
Plasma Cmax of PF-07304814 (prodrug) and PF 00835231 (active moiety) | 0-48 hours post the start of dosing
  Maximum plasma concentration
Plasma C24 of PF-07304814 (prodrug) and PF 00835231 (active moiety) | 0-48 hours post the start of dosing
  Plasma concentration at the end of infusion (24 hours post the start of infusion)
Plasma Css of PF-07304814 (prodrug) and PF 00835231 (active moiety) | 0-48 hours post the start of dosing
  Plasma steady state concertation
Plasma AUClast of PF-07304814 (prodrug) and PF 00835231 (active moiety) | 0-48 hours post the start of dosing
  Area under the serum concentration time profile from time zero to the time of the last quantifiable concentration.
Plasma AUCinf of PF-07304814 (prodrug) and PF 00835231 (active moiety) | 0-48 hours post the start of dosing
  Area under the serum concentration time profile from time zero to infinity.
Plasma AUCinf (dn) of PF-07304814 (prodrug) and PF 00835231 (active moiety) | 0-48 hours post the start of dosing
  Dose normalized AUCinf
Plasma Css (dn) of PF-07304814 (prodrug) and PF 00835231 (active moiety) | 0-48 hours post the start of dosing
  Dose normalized Css
Plasma t1/2 of PF-07304814 (prodrug) and PF 00835231 (active moiety) | 0-48 hours post the start of dosing
  Terminal half life
Plasma CL of PF-07304814 (prodrug) | 0-48 hours post the start of dosing
  Clearance
Plasma Vdss of PF-07304814 (prodrug) | 0-48 hours post the start of dosing
  Volume of distribution at steady state
PF-00835231 urinary PK: Ae | 0-36 hours post the start of dosing
  Amount of unchanged drug excreted in urine over collection interval
PF-00835231 urinary PK: Ae% | 0-36 hours post the start of dosing
  Percent of dose excreted in urine as unchanged drug over the collection interval.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- New Haven Clinical Research Unit, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- [Derived] Zhu T, Pawlak S, Toussi SS, Hackman F, Thompson K, Song W, Salageanu J, Winter E, Shi H, Winton J, Binks M. Safety, Tolerability, and Pharmacokinetics of Intravenous Doses of PF-07304814, a Phosphate Prodrug Protease Inhibitor for the Treatment of SARS-CoV-2, in Healthy Adult Participants. Clin Pharmacol Drug Dev. 2022 Dec;11(12):1382-1393. doi: 10.1002/cpdd.1174. Epub 2022 Oct 26. PMID 36285536
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C4611007